CLINICAL TRIAL: NCT02484118
Title: Examining the Effect of Blood Flow Rate on Hemodialysis Urea Clearance
Brief Title: Hemodialysis Blood Flow and Urea Clearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H14-01931
Record Dates: First submitted 2015-02-04; First posted 2015-06-29 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: End Stage Renal Failure on Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted blood flow rate 320 ml/min (Experimental): Hemodialysis blood flow will be targeted at 320 ml/min during hemodialysis for two weeks
  Interventions: Procedure: Hemodialysis blood flow
- Targeted blood flow rate 380 ml/min (Experimental): Hemodialysis blood flow will be targeted at 380 ml/min during hemodialysis for two weeks
  Interventions: Procedure: Hemodialysis blood flow

INTERVENTIONS:
Procedure: Hemodialysis blood flow — The impact of blood flow rates of 320 ml/m and 380 ml/m will be compared to determine any impact on hemodialysis urea clearance

SUMMARY:
The study purpose is to determine whether two different hemodialysis blood flow rates each meet national dialysis standards for urea clearance. Urea is used as the primary marker of dialysis adequacy. It is an experimental study with a crossover design of minimum 38 participants. Participants will be selected from the accessible pool of end-stage renal disease clients at the Vancouver Community Dialysis Unit. The participants will dialyse at each pre-determined blood flow rate (320 mL/min and 380 mL/min) for two weeks each. Two forms of urea clearance data will be collected: one value that is routinely calculated by the dialysis machine and recorded on client treatment logs, and another that is calculated in a lab from blood samples.

DETAILED DESCRIPTION:
Design This quasi-experimental study involves the independent variable of blood flow rate (Qb), measured in mL/min, and the dependent variable of dialysis clearance, measured by Kt/V and URR (urea reduction ratio). Control and randomization will be manifested in a crossover design, which provides the benefit of separating treatment effects from period effects (Wellek & Blettner, 2012). Participants will be randomly assigned - by way of selecting names from an envelope - to one of two groups: A, which dialyses first at 320 mL/min; or B, at 380 mL/min. Each study period will consist of two weeks (6 sessions, 24 hours of dialysis) at each Qb. Because urea clearance is immediate, six treatments at each Qb will reflect accurate data on Kt/V and URR (Dr. John Duncan, 2014, personal communication). Although carryover effects are not of concern to this study as participants routinely dialyse three times per week, wherein urea levels naturally rise between routine treatments, a washout phase of one week between study periods will occur, as is recommended for an effective crossover design (Wellek & Blettner, 2012).

Sample

The target and sample population are end-stage renal disease patients dialysing with an arteriovenous fistula (AVF) at the Vancouver Community Dialysis Unit. Power analysis was conducted by the Centre for Health Evaluation and Outcome Sciences (CHEOS). To ensure a Kt/V of 1.3 and URR of 70% can be estimated with a confidence interval of 95%, a minimum sample size of 34 participants is required. An additional 10% is necessary to account for attrition. Because randomization will occur with study period assignment, purposive sampling will be used to select participants from the accessible pool (estimated at 60 patients), until 38 participants are identified. The inclusion criteria are:

Dialysing for greater than six months to ensure access patency, viability, and stability; Undergoing thrice weekly, four-hour dialysis sessions for uniform dialysis duration; Dialysing with an AVF, either brachio-cephalic or radio-cephalic; no central venous catheters, arteriovenous grafts, or femoral AVFs due to differences in access flows and vessel quality; BLOOD FLOW RATE 5 Dialysing with 15g needles as organization policy restricts greater flow rates with smaller needle gauge; Dialysing with a dialysate flow (Qd) of 500 mL/min to reduce the possibility of clearance being attributable to differences in Qd; Maintaining transonic vascular access flows of >600 mL/min for the past 6 months, per KDOQI (NKF, 2006) minimum flow guidelines, to ensure access patency; Not part of any other research study that would interfere with dialysis treatment.

Data Collection Hourly documentation of Qb is routine protocol in the HD (hemodialysis) unit, along with Kt/V at each treatment termination. URR is routinely drawn every 6 weeks, however during this study it will be drawn weekly, on each third treatment. Standard URR blood draw protocol will be followed: a pre- and post- dialysis blood specimen will be collected and sent, along with the corresponding requisition, for analysis and calculation. A research account will be opened with LifeLabs (local laboratory service) and all research requisitions and blood will be coded and billed to the research study. Per unit protocol, blood draws will be written in the unit diary for nurse awareness, and blood collection tubes and requisition placed in participants' charts the night prior to treatment. Once weekly, the researchers will photocopy the participants' treatment run logs, along with the urea lab report, and data will be inputted into a CHEOS-approved excel spreadsheet. Along with Qb and Kt/V, collected data will include participants' blood pressure, dialysate flow rate, dialysis duration, needle gauge and cannulation, and occurrence of any intradialytic complications.

Data Analysis Data analysis will be conducted by CHEOS.

ELIGIBILITY:
Inclusion Criteria:

Participants will be selected from the Vancouver Community Dialysis Unit.

The inclusion criteria for participant selection will be:

1. Dialysing for greater than six months to ensure access patency, viability, and stability;
2. Undergoing thrice weekly, four-hour dialysis sessions for uniform dialysis duration;
3. Dialysing with an arteriovenous fistula, either brachio-cephalic or radio-cephalic, to control variances in blood flow rates related to vascular access;
4. Dialysing with 15g needles as organization policy restricts greater flow rates with smaller needle gauge;
5. Dialysing with a dialysate flow (Qd) of 500 mL/min to reduce the possibility of clearance being attributable to differences in Qd;
6. Maintaining transonic vascular access flows of >600 mL/min for the past 6 months, per Kidney Dialysis Outcomes Quality Initiative (KDOQI) (NKF, 2006) minimum flow guidelines, to ensure access patency.

Exclusion Criteria:

Patients who speak a language other than English, Cantonese, Mandarin, or Punjabi will be excluded due to funding constraints for providing translated informed consent documents. Informed consent documents will only be available in the languages listed above, which are the most common languages spoken/read at the dialysis unit.

Patients who dialyse with a central venous catheter, arteriovenous graft, or femoral arteriovenous fistula will not be invited to participate due to potential confounding from known differences in access flows and vessel quality that may impact clearance values.

Patients who are involved in any other research study that would interfere with their dialysis treatment would be excluded from the study.

Patients who are hemodynamically unstable (e.g.: frequent 'crashing' due to severe hypotension) will be excluded due to the instability this would pose on achieving their prescribed dialysis time (e.g.: if they crash, they may be taken off dialysis early) and resulting data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Urea clearance | Two weeks of dialysis at each blood flow rate

CONTACTS AND LOCATIONS:
Overall Officials: John A Duncan, MSc MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Division of Nephrology, Vancouver, British Columbia, Canada